CLINICAL TRIAL: NCT07136948
Title: Mindfulness Training and Respiration Biosignal Feedback - Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Equa Health (Industry)
Collaborators: Worcester Polytechnic Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Creswell, Co-Founder, Chief Science Officer, Equa Health
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R44MH134709-01A1 (NIH); 1R44MH134709-01A1 (NIH)
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Psychological Distress; Mindfulness Skills; Usability Satisfaction
Keywords: respiration biosignal feedback; young adults; mental health; well-being; mindfulness skills; psychological distress
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: The investigators will experimentally evaluate if Equa-augmented respiration biosignal tracking significantly increases user satisfaction relative to Equa with no biosignal tracking. Both groups will receive the 14 lessons of mindfulness meditation, however only one group (experimental) will see the respiration biosignal feedback from the algorithm developed and tested in Study 1.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group, No Physiological Feedback (Active Comparator): Participants be randomly assigned to one of two different 14-unit smartphone meditation program groups that involve completing a 2-10 minute daily guided practice on their phones. Participants in both groups will follow the same 14 units of mindfulness meditation curriculum that consists of learning and practicing techniques to improve concentration, sensory clarity, and equanimity (Equa meditation app) and have access to additional curriculum. Physiological measures will be tracked throughout the duration of lessons. A subset of participants (the experimental group) will see a graph tracking their physiological responses from the guided meditation lesson and predictive mindfulness skill scores based on the algorithm development. The control group will not see the graph tracking their physiology.
  Interventions: Behavioral: Mindfulness Meditation
- Experimental Group, Physiological Feedback (Experimental): Following the guided meditation lessons, a subset of participants (the experimental group) will see a graph tracking their physiological responses from the guided meditation lesson and predictive mindfulness skill scores based on the algorithm development. The feedback chart is produced by the physiological measures tracked throughout the duration of the lesson, and is displayed within the Equa app, moments after the meditation lessons concludes.
  Interventions: Behavioral: Mindfulness Meditation with Respiration Feedback Chart and Predictive Mindfulness Skill Scores

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Participants will be randomly assigned to one of two different 14-unit smartphone meditation program groups that involve completing a 2-10 minute daily guided practice on their phones. Participants in both groups will follow the same 14 units of mindfulness meditation curriculum that consists of learning and practicing techniques to improve concentration, sensory clarity, and equanimity (Equa meditation app) and have access to additional curriculum. Physiological measures will be tracked throughout the duration of lessons. The control group will not see the graph tracking their physiological responses or the predictive mindfulness skill scores based on the algorithm development.
  Arms: Control Group, No Physiological Feedback
Behavioral: Mindfulness Meditation with Respiration Feedback Chart and Predictive Mindfulness Skill Scores — Participants will then be randomly assigned to one of two different 14-unit smartphone meditation program groups that involve completing a 2-10 minute daily guided practice on their phones. Participants in both groups will follow the same 14 units of mindfulness meditation curriculum that consists of learning and practicing techniques to improve concentration, sensory clarity, and equanimity (Equa meditation app) and have access to additional curriculum. Physiological measures will be tracked throughout the duration of lessons. Following the guided meditation lessons, a subset of participants (the experimental group) will see a graph tracking their physiological responses from the guided meditation lesson and predictive mindfulness skill scores based on our algorithm development. The feedback chart is produced by the physiological measures tracked throughout the duration of the lesson, and is displayed within the Equa app, moments after the meditation lessons concludes.
  Arms: Experimental Group, Physiological Feedback

SUMMARY:
The goal of this research is to test usability and user satisfaction with a new breathing feature on the meditation app, Equa, to help young adults who are distressed, understand their physiological responses and mindfulness skill development during meditation.

Our main aims are to test an algorithm that can use physiologic signals to give feedback about how participant physiology is changing during guided lessons on the meditation app, Equa through:

* Assessing user satisfaction and usability
* Measuring how much participant mindfulness skills are improving

Participants will:

* Complete a survey about demographics, their thoughts and feelings before and after the mindfulness meditation program
* Complete 14 smartphone guided mindfulness meditation training units while physiological measures are being recorded
* A subset of participants will see a graph tracking their physiological responses from the guided meditation lesson and predictive mindfulness skill scores
* Complete a few brief questionnaires before and after mindfulness practices to understand potential changes in their mindfulness skills

DETAILED DESCRIPTION:
Investigators will recruit young adults to participate in a study to examine the usability and user satisfaction of respiration biosignal feedback during meditation through phone motion data and microphones within headphones. Interested participants will be screened on study inclusion/exclusion criteria: (1) aged 18-30 years, (2) interested in coming on site to complete 14 smartphone guided mindfulness meditation training units, (3) willing to be assigned to one of two conditions, (4) willing to wear physiological monitoring equipment and provide ratings of their training experience, (5) Not currently pregnant and (6) no current or previous diagnosis of psychosis or schizophrenia

Participants are told they are going to participate in a study that focuses on monitoring physiological responses during meditation. At the start of the study, participants will complete questions via an online survey focused on demographics, prior meditation experience, their thoughts and feelings as these may be informative to participants' meditation experience.

Participants will complete a few brief questionnaires to understand potential changes in mindfulness before and after select lessons. Participant physiological data will be recorded (E.g., heart rate) via smartphones and headphones to track physiologic dynamics. Additionally, the sensory shirt, made by Hexoskin Smart Sensors; AI, will also continuously measure physiologics via two inductive plethysmography (RIP) sensors. The Hexoskin shirt also tracks motion via a three-axis accelerometer. These measures will enable investigators to better understand mindfulness measures during meditation.

Following the guided meditation lessons, a subset of participants (the experimental group) will see a graph tracking their physiological responses from the guided meditation lesson and predictive mindfulness skill scores based on our algorithm development. The feedback chart is produced by the physiological measures tracked throughout the duration of the lesson, and is displayed within the Equa app, moments after the meditation lessons concludes. The control group will not see the graph tracking their physiological responses.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30 years of Age
* Fluent in English
* Psychological distress
* Willing to participate in guided meditation or stress management training.
* Willing and able to wear earbud headphones and a shirt which uses sensors to track motion and physiological measures.
* Willing to be randomized to one of two conditions
* Willing to provide ratings on their training experience

Exclusion Criteria:

* Currently pregnant
* Current or previous diagnosis with psychosis or schizophrenia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Assess usability and user satisfaction with respiration biosignal tracking and predictive mindfulness skill scores during meditation training to changes in mindfulness skills from pre-training to post-training | Throughout 5 sessions over the course of 4 weeks (study completion)
  >85 on System Usability Scale and significantly more user satisfaction with biosignal augmented Equa.
  The investigators will conduct usability testing with the respiration biosignal tracking on Equa, and experimentally evaluate if Equa-augmented respiration biosignal tracking increases user satisfaction in the lab relative to Equa with no biosignal tracking.

SECONDARY OUTCOMES:
Change from Baseline in total anxiety as assessed by the General Anxiety Disorder, 7-item questionnaire at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking about how often they have been bothered by any of the listed problems over the last 2 weeks. Zero is equivalent to not at all (lower anxiety) and 3 indicates nearly every day (higher anxiety).
Change from Baseline in total depression as assessed by the Patient Health Questionnaire-9 at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking about how often they have been bothered by any of the listed problems over the last 2 weeks related to the severity of depression symptomology. Zero is equivalent to not at all (lower depression) and 3 indicates nearly every day (higher depression)
Change from Baseline in total affect as assessed by the Positive and Negative Affect Scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking to indicate the extent they have felt the following ways over the past 2 weeks related to their feelings and emotions. One is equivalent to not at all and five indicates extremely. The scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19 are added. Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. The scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20 are added. Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Change from Baseline in mean state mindfulness as assessed by the Mindful Attention Awareness Scale - state at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking to what degree they were having each experience described over the past 2 weeks related to mindfulness practices. Zero is equivalent to not at all and six indicates very much. A mean score of the 15 items is taken, a higher score indicates greater mindfulness and a lower score indicates lower mindfulness.
Change from Baseline in total perceived stress as assessed by the Perceived Stress Scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking about their feelings and thoughts over the past 2 weeks. Zero is equivalent to never and four indicates very often. Scores are added and those ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress and scores ranging from 27-40 would be considered high perceived stress.
Change from Baseline in total social well-being as assessed by the Satisfaction with Life Scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. A score of 5-9 indicates extreme dissatisfaction and a score of 31-35 indicates extreme satisfaction.
Change from Baseline in total loneliness as assessed by the UCLA Loneliness scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants indicate how often they feel the way related to loneliness and isolation described in each of the 20 statements using a 4-point scale that ranges from 1=never to 4=always. The scoring is continuous with items 1, 5, 6, 9, 10, 15, 16, 19, 20 are all reverse scored. A higher score indicates greater feelings of isolation and loneliness, while a lower score indicates lower feelings of isolation and loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: David Creswell, Ph.D., Principal Investigator — Equa Health
Locations (1):
- GATF Building, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will only share de-identified data from our studies that allows outside groups to independently validate our claims in our published scientific articles. All data and documentation will be de-identified and will be consistent with applicable laws and regulations.
Supporting Information: Study Protocol, ICF
Time Frame: The investigators will provide data within six months of any approved request.
Access Criteria: Scientific groups who aim to validate our findings can make requests for data access. The study team agrees that the names and Institutions of persons either given or denied access to the data, and the bases for such decisions, will be summarized in the annual progress reports.